CLINICAL TRIAL: NCT02161692
Title: Randomized Phase 2 Study of Conventional Dose Chemotherapy Versus High Dose Sequential Chemotherapy as First-line Therapy for Metastatic Poor Prognosis Germ Cell Tumors
Brief Title: Conventional Dose Versus High Dose Sequential Chemotherapy for Poor Prognosis Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Andrea Necchi, Faculty, Department of Medical Oncology, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT48/96
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Testicular Neoplasms; Germ Cell Tumors
MeSH Terms: conditions — Testicular Neoplasms; Neoplasms, Germ Cell and Embryonal | interventions — Cyclophosphamide; Etoposide; Cisplatin; Bleomycin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose chemotherapy (Experimental): Characterized by the following sequence:
  High dose cyclophosphamide (7 grams/squared meter) x 1 cycle 2 cycles of high-dose etoposide and cisplatin
  1 cycle of high dose carboplatin (Area Under the Curve 27) with stem cell rescue
  Interventions: Drug: Cyclophosphamide; Drug: Etoposide; Drug: Cisplatin; Drug: Carboplatin
- Conventional dose chemotherapy (Active Comparator): Cisplatin, Etoposide, and Bleomycin (PEB) x 4 cycles
  Interventions: Drug: Etoposide; Drug: Cisplatin; Drug: Bleomycin

INTERVENTIONS:
Drug: Cyclophosphamide
  Arms: High dose chemotherapy
Drug: Etoposide
Drug: Cisplatin
Drug: Bleomycin
  Arms: Conventional dose chemotherapy
Drug: Carboplatin — High dose carboplatin
  Arms: High dose chemotherapy

SUMMARY:
The purpose of this study is to determine whether the use of a sequential high dose chemotherapy is more effective than conventional dose (i.e. 4 cycles of cisplatin, etoposide, and bleomycin [PEB]) in patients with metastatic poor prognosis germ cell tumors.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or Histological diagnosis of germ cell tumors
* Metastatic disease
* Poor prognostic category according to the International Germ Cell Collaborative Group (IGCCCG) classification
* No prior chemotherapy for metastatic disease

Exclusion Criteria:

* Unwillingness to accomplish the study procedures
* Any existing co-morbidity that could limit the administration of high dose chemotherapy
* Any psychiatric disorder that could impact on the study compliance

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-12; Primary Completion 2007-05 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Evidence of disease progression confirmed by computed tomography (CT) scan and/or serum tumor markers. | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Necchi, MD, Principal Investigator — Istituto Nazionale dei Tumori, Milano Italy
Locations (1):
- Istituto Nazionale dei Tumori, Milan, Milano, Italy

REFERENCES:
- [Background] Lorch A, Bascoul-Mollevi C, Kramar A, Einhorn L, Necchi A, Massard C, De Giorgi U, Flechon A, Margolin K, Lotz JP, Germa-Lluch JR, Powles T, Kollmannsberger C, Beyer J. Conventional-dose versus high-dose chemotherapy as first salvage treatment in male patients with metastatic germ cell tumors: evidence from a large international database. J Clin Oncol. 2011 Jun 1;29(16):2178-84. doi: 10.1200/JCO.2010.32.6678. Epub 2011 Mar 28. PMID 21444870
- [Derived] Necchi A, Mariani L, Di Nicola M, Lo Vullo S, Nicolai N, Giannatempo P, Raggi D, Fare E, Magni M, Piva L, Matteucci P, Catanzaro M, Biasoni D, Torelli T, Stagni S, Bengala C, Barone C, Schiavetto I, Siena S, Carlo-Stella C, Pizzocaro G, Salvioni R, Gianni AM. High-dose sequential chemotherapy (HDS) versus PEB chemotherapy as first-line treatment of patients with poor prognosis germ-cell tumors: mature results of an Italian randomized phase II study. Ann Oncol. 2015 Jan;26(1):167-172. doi: 10.1093/annonc/mdu485. Epub 2014 Oct 24. PMID 25344361